CLINICAL TRIAL: NCT06615882
Title: An Exploratory Study of Intra-arterial Mechanical Angioplasty Using a SOLITAIRE™ X Stent for Refractory and Recurrent Vasospasm Mechanical Intracranial Artery DilAtation Using Stent-retriever for Cerebral Vasospasm
Brief Title: Mechanical Intracranial Artery DilAtation Using Stent-retriever for Cerebral Vasospasm
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-2024-0013
Record Dates: First submitted 2024-09-08; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Intracranial Vasospasm
MeSH Terms: conditions — Vasospasm, Intracranial | interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): During the stent (Solitaire-X) -angioplasty, IA nimodipine was also infused
  Interventions: Device: stent-angioplasty & nimodipine infusion (During the stent (Solitaire-X) -angioplasty, IA nimodipine was also infused)

INTERVENTIONS:
Device: stent-angioplasty & nimodipine infusion (During the stent (Solitaire-X) -angioplasty, IA nimodipine was also infused) — I. Procedure & Intervention
  1. Assess the presence and degree of cerebral vasospasm of the target vessel through cerebral angiography before the procedure.
  2. Solitaire-X stent types are selected
  3. During the stent-angioplasty, IA nimodipine was also infused.
  4. Retrieve Solitaire-X after maintaining deployment for 3 minutes.
  5. Additional procedures are determined through immediate post-procedure and 15-minute delayed cerebral angiography.

SUMMARY:
Solitaire-x is a stent-retriever that is currently world-widely used, but is currently FDA-approved only as a revascularization device indicated for use to restore blood flow in the neurovasculature by removing thrombus for the treatment of acute ischemic stroke. Its utility for mechanical endovascular dilatation for refractory intracranial vasospasm is an off-label indication. In this reason, we designed single-arm, prospective study, which aimed to report the safety and effectiveness of Solitaire-X in CV after subarachnoid Prospective exploratory study, single arm (off label), single center study

DETAILED DESCRIPTION:
Prospective exploratory study, single arm (off label), single center study I. Procedure & Intervention

1. Assess the presence and degree of cerebral vasospasm of the target vessel through cerebral angiography before the procedure.
2. Solitaire-X stent types are selected
3. During the stent-angioplasty, IA nimodipine was also infused.
4. Retrieve Solitaire-X after maintaining deployment for 3 minutes.
5. Additional procedures are determined through immediate post-procedure and 15-minute delayed cerebral angiography.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients≥ 19 years 2. Radiologic confirmed refractory intracranial vasospasm or due to subarachnoid hemorrhage (caused by trauma, aneurysmal rupture, spontaneous, etc.) or suspected recurrent intracrania vasospasm with the following radiological/clinical evidence (* refractory intracranial vasospasm: despite of standard treatment ≥ 50% decrease in vessel diameter compared to first angiography)

  * recurrent intracrania vasospasm: Even though chemical angioplasty was performed, radiologically cerebral vasospasm worsens (severe cerebral vasospasm(70-99%)) with worsening clinical symptoms.

    3. Individuals who voluntarily signed the informed consent form to participate in this study.

Exclusion Criteria:

* 1. Pre-existing intracranial stenosis ≥ 50% 2. Patients whose condition makes further evaluation and procedures difficult
* Exclude if Hunt and Hess grade is 4 or higher. 3. Difficult vascular access
* History of vascular malformation, vascular anastomosis, or stent placement. 4. Distal location: Middle cerebral artery (MCA) segment M3 or below, anterior cerebral artery (ACA) segment A3 or below, posterior cerebral artery (PCA) segments P3 or P4 or below.

  5. Cerebral vasospasm caused by vasculitis or dissection. 6. Hypersensitivity to medications to be used (contrast agents, vasodilators..).

  7. Pregnancy or breastfeeding. 8. History of connective tissue disease or blood coagulation disorders. 9. Patients with untreated areas of subarachnoid hemorrhage. 10. Patients with symptoms due to other causes (e.g., hydrocephalus, infection, etc.).

  11. Irreversible cerebral infarction in the entire vascular territory where vasospasm occurred.

  12. Known allergy to medical device materials (Nitinol, Platinum, Iridium). 13. Bleeding or coagulation disorders (Platelet count < 20,000 or INR > 1.7). 14. In case of rapid worsening of cerebral hemorrhage symptoms , cerebral edema, surgery, or other urgent treatment required.

  15. Subject with uncontrolled blood pressure (SBP < 100 mmHg). 16. Subject with liver dysfunction (AST/ALT > x2 upper normal limit ). 17. Subject with renal dysfunction (eGFR < 60 mL/min/1.73㎡). 18. Subject with clinically significant cardiac complications such as arrhythmia, heart failure, or myocardial infarction.

  19. Subject with brain edema or elevated intracranial pressure. 20. Known current or past use of illicit drugs or alcohol abuse. 21. Requiring the administration of medications contraindicated with nimodipine.

  22. Subject with systemic complications such as infection, fever, inflammation, edema, hypersensitivity, foreign body reaction, toxicity, or shock.

  23. Subject with visual impairment or ocular complications. 24. Any other cases where the investigator determines that participation in the clinical trial is not possible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Assess the safety (adverse events) of the interventional procedure. | at 24 hours and 72 hours after the intervention at 3 months after Cerebral Vasospasm Onset.

SECONDARY OUTCOMES:
Intervention Success Rate | at 24 hours and 72 hours after the intervention at 3 months after Cerebral Vasospasm Onset.
  Recovery of more than 50% of the pre-procedure vessel diameter, measured at 24 hours and 72 hours after the intervention.
Whether additional treatment is required after intervention (; in relation to cerebral vasospasm) questionnaire | On the 1 day of the subject's intervention
Symptom Improvement (NIHSS) | Improvement in NIHSS at 3 months after Cerebral Vasospasm Onset.
  NIHSS: National Institutes of Health Stroke Scale Score 0: no stroke Score 1-4: minor stroke Score 5-15: moderate stroke Score 15-20: moderate to severe stroke Score 21-42: severe stroke
Clinical Improvement (mRS) | at 24 hours and 72 hours after the intervention at 3 months after Cerebral Vasospasm Onset.
  mRS: Modified Rankin Score 0: None
  1. No significant disability despite symptoms: able to carry out all usual duties and activities
  2. Slight disability: unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability: requiring some help, but able to walk without assistance
  4. Moderately severe disability: unable to walk without assistance, unable to attend to needs without assistance
  5. Severe disability: bed-ridden, incontinent, and requiring constant nursing care and attention
  6. Dead
Degree of Cerebral Vasospasm | observed in CT cerebral angiography at 24 hours and 72 hours after the intervention.
  * Visual classification: Cerebral vasospasm grades (CVSG). Grade 0 All intracranial vessels show a physiological shape Grade 1 Vasospasm affects the A2, A1, and M2 segments Grade 2 Vasospasm expands to the M1 and terminal segment of the internal carotid artery Grade 3 Severe reduction in the intradural internal carotid artery with filiform A1 and M1 segments, which sometimes appears like a ghost (ghost sign)
  * Degree of diameter reduction
    * None (0-10%),
    * Mild (11-49%),
    * Moderate (50-69%),
    * Severe (70-99%)

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei university college of medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No